CLINICAL TRIAL: NCT00381641
Title: Phase II Trial of Sunitinib (SU11248) in Iodine-131 Refractory, Unresectable Differentiated Thyroid Cancers and Medullary Thyroid Cancers
Brief Title: Sunitinib Malate in Treating Patients With Thyroid Cancer That Did Not Respond to Iodine I 131 and Cannot Be Removed by Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00213; NCI-2009-00213 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); UCCRC-14696A; CDR0000502260; NCI-7735; 14696A; 7735 (Other: University of Chicago Comprehensive Cancer Center); 7735 (Other: CTEP); N01CM62201 (NIH); N01CM62202 (NIH); P30CA014599 (NIH)
Record Dates: First submitted 2006-09-26; First posted 2006-09-28 (Estimated); Results first posted 2017-09-15 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Differentiated Thyroid Gland Carcinoma; Recurrent Thyroid Gland Carcinoma; Refractory Thyroid Gland Carcinoma; Stage III Thyroid Gland Follicular Carcinoma AJCC v7; Stage III Thyroid Gland Medullary Carcinoma AJCC v7; Stage IV Thyroid Gland Follicular Carcinoma AJCC v7; Stage IV Thyroid Gland Medullary Carcinoma AJCC v7; Stage IV Thyroid Gland Papillary Carcinoma AJCC v7; Stage IVA Thyroid Gland Follicular Carcinoma AJCC v7; Stage IVA Thyroid Gland Medullary Carcinoma AJCC v7; Stage IVA Thyroid Gland Papillary Carcinoma AJCC v7; Stage IVB Thyroid Gland Follicular Carcinoma AJCC v7; Stage IVB Thyroid Gland Medullary Carcinoma AJCC v7; Stage IVB Thyroid Gland Papillary Carcinoma AJCC v7; Stage IVC Thyroid Gland Follicular Carcinoma AJCC v7; Stage IVC Thyroid Gland Medullary Carcinoma AJCC v7; Stage IVC Thyroid Gland Papillary Carcinoma AJCC v7; Thyroid Gland Oncocytic Carcinoma; Unresectable Thyroid Gland Carcinoma
MeSH Terms: conditions — Thyroid Neoplasms; Adenocarcinoma, Follicular; Carcinoma, Medullary; Thyroid Cancer, Papillary | interventions — Pharmacogenomic Testing; Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (sunitinib malate) (Experimental): Patients receive sunitinib malate PO QD on days 1-28. Cycles repeat every 6 weeks in the absence of disease progression or unacceptable toxicity
  Interventions: Other: Laboratory Biomarker Analysis; Other: Pharmacogenomic Study; Drug: Sunitinib; Drug: Sunitinib Malate

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Optional correlative studies
Other: Pharmacogenomic Study — Optional correlative studies
  Other Names: PHARMACOGENOMIC
Drug: Sunitinib — Given PO
Drug: Sunitinib Malate — Given PO
  Other Names: SU 011248; SU 11248; SU-011248; SU-11248; SU011248; SU11248; sunitinib; Sutent

SUMMARY:
This phase II trial studies how well sunitinib malate works in treating patients with thyroid cancer that did not respond to iodine I 131 (radioactive iodine) and cannot be removed by surgery. Sunitinib malate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the response rate of single agent sunitinib (sunitinib malate) in patients with iodine refractory, unresectable well-differentiated thyroid cancer (WDTC) who have evidence of disease progression within 6 months of study enrollment.

II. Determine the response rate of single agent sunitinib in patients with medullary thyroid cancer (MTC) who have evidence of disease progression within 6 months of study enrollment.

III. Determine the toxicity, duration of response, progression free survival, and overall survival in patients with WDTC or MTC treated with single agent sunitinib.

IV. Determine whether the presence of ret proto-oncogene (RET) gene rearrangements in patients with WDTC or RET mutations in patients with MTC predict response to sunitinib.

V. Determine whether therapy with sunitinib affects phosphorylation of downstream RET effector, mitogen-activated protein kinase 1 (ERK), in WDTC and MTC tissue.

VI. Determine whether specific germ-line polymorphisms in the RET gene are associated with favorable outcome in patients with WDTC treated with sunitinib.

OUTLINE: Patients are assigned to 1 of 2 cohorts according to type of thyroid cancer (medullary vs well-differentiated).

Patients receive sunitinib malate orally (PO) once daily (QD) on days 1-28. Cycles repeat every 6 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up periodically for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed papillary, follicular, or Hurthle cell carcinoma (cohort A) or medullary thyroid carcinoma (cohort B); their disease must have progressed despite treatment with iodine-131 therapy or they are not candidates for iodine-131 therapy and their disease cannot be completely removed by surgery; all patients with WDTC are expected to be on thyroxine suppression therapy
* Patients must have radiographically or biochemically measurable disease; radiographically measurable disease is defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as >= 20 mm with conventional techniques or as >= 10 mm with spiral computed tomography (CT) scan; biochemically measurable disease is defined as an elevated thyroglobulin (WDTC patients) or calcitonin (MTC patients)
* Patients must have evidence of disease progression (objective growth of existing tumors or rising thyroglobulin or calcitonin levels) within the last 6 months
* Patients cannot have received prior receptor tyrosine kinase inhibitors; patients cannot have received more than one prior chemotherapy regimen for metastatic disease; patients cannot have received prior external beam radiation to the measured tumor constituting the target lesion(s)
* Life expectancy of greater than 12 weeks
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2 (Karnofsky >= 60%)
* Leukocytes >= 3,000/mcL
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Hemoglobin >= 9 g/dL
* Serum calcium =< 12.0 mg/dL
* Total serum bilirubin within normal institutional limits
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 X institutional upper limit of normal OR =< 5 X institutional upper limit of normal if patient has liver metastases
* Creatinine within normal institutional limits OR creatinine clearance >= 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* Patients must have corrected QT interval (QTc) < 500 msec
* The following groups of patients are eligible provided they have New York Heart Association class II (NYHA) cardiac function on baseline echocardiogram (ECHO)/multigated acquisition scan (MUGA):

  * Those with a history of class II heart failure who are asymptomatic on treatment
  * Those with prior anthracycline exposure
  * Those who have received central thoracic radiation that included the heart in the radiotherapy port
* The effects of sunitinib on the developing human fetus at the recommended therapeutic dose are unknown; for this reason and because antiangiogenic agents are known to be teratogenic, women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; all women of childbearing potential must have a negative pregnancy test prior to receiving sunitinib; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier; at least 4 weeks must have elapsed since any major surgery
* Patients may not be receiving any other investigational agents
* Patients who have received prior treatment with any other antiangiogenic agent (e.g., bevacizumab, sorafenib, pazopanib, AZD2171, PTK787, vascular endothelial growth factor [VEGF] Trap, etc.)
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to sunitinib
* Patients with QTc prolongation (defined as a QTc interval equal to or greater than 500 msec), serious ventricular arrhythmia (ventricular fibrillation or ventricular tachycardia greater than or equal to 3 beats in a row) or other significant electrocardiogram (ECG) abnormalities are excluded
* Patients with poorly controlled hypertension (systolic blood pressure of 140 mmHg or higher or diastolic blood pressure of 90 mmHg or higher) are ineligible
* Patients who require use of therapeutic doses of coumarin-derivative anticoagulants such as warfarin are excluded, although doses of up to 2 mg daily are permitted for prophylaxis of thrombosis; Note: Low molecular weight heparin is permitted provided the patient's prothrombin time (PT) international normalized ratio (INR) is =< 1.5
* Patients with any condition (e.g., gastrointestinal tract disease resulting in an inability to take oral medication or a requirement for intravenous [IV] alimentation, prior surgical procedures affecting absorption, or active peptic ulcer disease) that impairs their ability to swallow and retain sunitinib tablets are excluded
* Patients with any of the following conditions are excluded:

  * Serious or non-healing wound, ulcer, or bone fracture
  * History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 28 days of treatment
  * Any history of cerebrovascular accident (CVA) or transient ischemic attack within 12 months prior to study entry
  * History of myocardial infarction, cardiac arrhythmia, stable/unstable angina, symptomatic congestive heart failure, or coronary/peripheral artery bypass graft or stenting within 12 months prior to study entry
  * History of pulmonary embolism within the past 12 months
  * Class III or IV heart failure as defined by the NYHA functional classification system
* Because sunitinib is metabolized primarily by the CYP3A4 liver enzyme, the eligibility of patients taking medications that are potent inducers or inhibitors of that enzyme will be determined following a review of their case by the principal investigator; every effort should be made to switch patients taking such agents or substances to other medications, particularly patients with gliomas or brain metastases who are taking enzyme-inducing anticonvulsant agents
* Patients with known brain metastases should be excluded because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events; N.B.: Patients with brain metastases with stable neurologic status following local therapy (surgery or radiation) for at least 8 weeks from definitive therapy and without neurologic dysfunction that would confound the evaluation of neurologic and other adverse events are eligible for participation; patients cannot be receiving enzyme inducing anti-convulsants including carbamazepine, phenobarbital, and phenytoin
* Patients with uncontrolled intercurrent illness including, but not limited to, ongoing or active infections or psychiatric illness/social situations that would limit compliance with study requirements are ineligible
* Pregnant women are excluded from this study because sunitinib is an antiangiogenic agent with the potential for teratogenic or abortifacient effects; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with sunitinib, breastfeeding should be discontinued if the mother is treated with sunitinib malate
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with sunitinib; in addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy; appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated
* Patients with conditions classified as NYHA III or IV per the New York Heart Association classifications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2006-08-29 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2024-12-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tanguy Y Seiwert, Principal Investigator — University of Chicago Comprehensive Cancer Center
Locations (17):
- United States (17):
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Duly Health and Care Joliet, Joliet, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Central Illinois Hematology Oncology Center, Springfield, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Fort Wayne Medical Oncology and Hematology Inc-Parkview, Fort Wayne, Indiana
  - Northern Indiana Cancer Research Consortium, South Bend, Indiana
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Oncology Care Associates PLLC, Saint Joseph, Michigan
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - M D Anderson Cancer Center, Houston, Texas
  - Medical College of Wisconsin, Milwaukee, Wisconsin

RESULTS

PARTICIPANT FLOW:
Groups:
- Sunitinib Malate-Radioactive Iodine Refractory Subgroup: Patients receive sunitinib malate PO QD on days 1-28. Courses repeat every 6 weeks in the absence of disease progression or unacceptable toxicity
  This arm contains results for the Radioactive Iodine Refractory Thyroid Cancer Subgroup
  Sunitinib Malate: Given PO
- Sunitinib Malate-Metastatic Medullary Subgroup: Patients receive sunitinib malate PO QD on days 1-28. Courses repeat every 6 weeks in the absence of disease progression or unacceptable toxicity
  This arm contains results for the Metastatic Medullary Thyroid Cancer Subgroup
  Sunitinib Malate: Given PO
Period: Overall Study
Arm/Group | Sunitinib Malate-Radioactive Iodine Refractory Subgroup | Sunitinib Malate-Metastatic Medullary Subgroup
Started | 38 | 25
Completed | 38 | 23
Not Completed | 0 | 2
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sunitinib Malate-Radioactive Iodine Refractory Subgroup | Sunitinib Malate-Metastatic Medullary Subgroup | Total
Number analyzed (Participants) | 38 | 25 | 63
Age, Continuous [Mean (Full Range); unit: years] | 59.1 [37 to 76] | 50.9 [23 to 73] | 55.8 [23 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 12 | 26
  Male | 24 | 13 | 37
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 4 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 37 | 20 | 57
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 38 | 25 | 63

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate, Assessed Using the Response Evaluation Criteria in Solid Tumors (RECIST)
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by CT or MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR."
Time Frame: Up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Sunitinib Malate-Radioactive Iodine Refractory Subgroup | Sunitinib Malate-Metastatic Medullary Subgroup
Number analyzed (Participants) | 38 | 25
Participants | 9 | 7
Statistical Analysis 1: Comparison: Sunitinib Malate-Radioactive Iodine Refractory Subgroup vs Sunitinib Malate-Metastatic Medullary Subgroup; Note. The objective was not to compare the two arms (subgroups), but to compare each with historical data; Test type: Superiority — Null (historical) response rate for iodine refractory subgroup is 10%. Power=90% for 30% alternative. Null (historical) response rate for metastatic medullary subgroup is 5%. Power=88% for 25% alternative; p < 0.10, Simon, two-stage design — For iodine refractory subgroup, null hypothesis could be rejected if 6 or more responses were observed. For metastatic medullary subgroup, null hypothesis could be rejected if 3 or more responses were observed

2. Secondary Outcome: Incidence of Toxicity, Graded According to the Common Terminology Criteria for Adverse Events Version 3.0
Description: Any grade toxicity of any type, regardless of attribution
Time Frame: From time of first treatment with sunitinib, assessed up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Sunitinib Malate-Radioactive Iodine Refractory Subgroup | Sunitinib Malate-Metastatic Medullary Subgroup
Number analyzed (Participants) | 38 | 25
Participants | 38 | 24

3. Secondary Outcome: Overall Survival
Description: Kaplan-Meier curves will be generated and 95% confidence intervals will be derived for median overall survival.
Time Frame: Up to 10 years
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Sunitinib Malate-Radioactive Iodine Refractory Subgroup | Sunitinib Malate-Metastatic Medullary Subgroup
Number analyzed (Participants) | 38 | 25
Months | 32.6 [18.4 to 70.9] | 65.4 [27.0 to 69.5]

4. Secondary Outcome: Time to Progression or Death Evaluated Using the RECIST
Time Frame: Time from start of treatment to time of progression or death of any cause, assessed up to 10 years
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Sunitinib Malate-Radioactive Iodine Refractory Subgroup | Sunitinib Malate-Metastatic Medullary Subgroup
Number analyzed (Participants) | 38 | 25
Months | 12.8 [8.3 to 16.4] | 19.3 [7.7 to 34.6]

5. Other Pre Specified Outcome: Changes in Laboratory Correlates Analyzed Using Paired T-tests
Description: Relevant laboratory correlates will be compared between responders and non-responders using the Wilcoxon rank sum test. The association between the presence or absence of RET gene rearrangements/mutations and tumor response, as well as the association between germ-line polymorphisms in the RET gene and response, will be analyzed using Fisher's exact test. The correlative and genetic data will also be entered as covariates (univariate analyses only due to the small sample size) in a Cox regression model of progression-free survival.
Time Frame: Baseline to 2 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Sunitinib Malate-Radioactive Iodine Refractory Subgroup | Sunitinib Malate-Metastatic Medullary Subgroup
All-Cause Mortality (participants affected / at risk) | 21/38 | 5/25
Serious Adverse Events (participants affected / at risk) | 17/38 | 12/25
Other Adverse Events (participants affected / at risk) | 38/38 | 24/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sunitinib Malate-Radioactive Iodine Refractory Subgroup (N=38) | Sunitinib Malate-Metastatic Medullary Subgroup (N=25)
Abdominal pain (Gastrointestinal disorders) | 0 | 2
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Buttock pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Cardiac disorders - Other (Cardiac disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Death NOS (General disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Fatigue (General disorders) | 1 | 0
Gastric hemorrhage (Gastrointestinal disorders) | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 2 | 0
Hypertension (Vascular disorders) | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 1 | 0
Infections and infestations - Other (Infections and infestations) | 0 | 1
Laryngeal edema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Laryngeal obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Left ventricular systolic dysfunction (Cardiac disorders) | 2 | 0
Mucositis oral (Gastrointestinal disorders) | 0 | 1
Neutrophil count decreased (Investigations) | 1 | 0
Oral pain (Gastrointestinal disorders) | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 1
Peripheral motor neuropathy (Nervous system disorders) | 0 | 1
Platelet count decreased (Investigations) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Reproductive system and breast disorders - Other (Reproductive system and breast disorders) | 0 | 1
Skin infection (Infections and infestations) | 1 | 0
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Tracheal fistula (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sunitinib Malate-Radioactive Iodine Refractory Subgroup (N=38) | Sunitinib Malate-Metastatic Medullary Subgroup (N=25)
Abdominal pain (Gastrointestinal disorders) | 4 | 5
Alanine aminotransferase increased (Investigations) | 14 | 6
Alkaline phosphatase increased (Investigations) | 8 | 4
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 7
Anemia (Blood and lymphatic system disorders) | 29 | 14
Anorexia (Metabolism and nutrition disorders) | 13 | 9
Anxiety (Psychiatric disorders) | 3 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 4
Aspartate aminotransferase increased (Investigations) | 16 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 6
Blood bilirubin increased (Investigations) | 3 | 4
Bone pain (Musculoskeletal and connective tissue disorders) | 3 | 0
Bronchial infection (Infections and infestations) | 2 | 0
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Bruising (Injury, poisoning and procedural complications) | 0 | 2
Constipation (Gastrointestinal disorders) | 13 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 10 | 4
Creatinine increased (Investigations) | 6 | 1
Dehydration (Metabolism and nutrition disorders) | 2 | 1
Diarrhea (Gastrointestinal disorders) | 25 | 11
Dizziness (Nervous system disorders) | 5 | 4
Dry mouth (Gastrointestinal disorders) | 5 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 5 | 1
Dysgeusia (Nervous system disorders) | 10 | 6
Dyspepsia (Gastrointestinal disorders) | 14 | 1
Dysphagia (Gastrointestinal disorders) | 2 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 7 | 3
Edema face (General disorders) | 2 | 8
Edema limbs (General disorders) | 4 | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 8 | 4
Eye disorders - Other (Eye disorders) | 0 | 2
Fatigue (General disorders) | 33 | 18
Fever (General disorders) | 6 | 2
Flatulence (Gastrointestinal disorders) | 2 | 1
Gastritis (Gastrointestinal disorders) | 3 | 2
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 2 | 2
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 3
Headache (Nervous system disorders) | 9 | 6
Hot flashes (Vascular disorders) | 3 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 27 | 17
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 3
Hypernatremia (Metabolism and nutrition disorders) | 2 | 2
Hypertension (Vascular disorders) | 18 | 4
Hyperthyroidism (Endocrine disorders) | 0 | 4
Hypoalbuminemia (Metabolism and nutrition disorders) | 10 | 3
Hypocalcemia (Metabolism and nutrition disorders) | 12 | 10
Hypoglycemia (Metabolism and nutrition disorders) | 4 | 1
Hypokalemia (Metabolism and nutrition disorders) | 7 | 4
Hyponatremia (Metabolism and nutrition disorders) | 4 | 3
Hypophosphatemia (Metabolism and nutrition disorders) | 6 | 4
Hypotension (Vascular disorders) | 2 | 0
Hypothyroidism (Endocrine disorders) | 1 | 4
Insomnia (Psychiatric disorders) | 4 | 1
Investigations - Other (Investigations) | 0 | 6
Lipase increased (Investigations) | 0 | 3
Lung infection (Infections and infestations) | 2 | 1
Lymphocyte count decreased (Investigations) | 20 | 14
Mucositis oral (Gastrointestinal disorders) | 18 | 12
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 3
Nail loss (Skin and subcutaneous tissue disorders) | 1 | 2
Nausea (Gastrointestinal disorders) | 20 | 13
Neck pain (Musculoskeletal and connective tissue disorders) | 3 | 0
Neutrophil count decreased (Investigations) | 21 | 8
Non-cardiac chest pain (General disorders) | 3 | 2
Oral pain (Gastrointestinal disorders) | 5 | 2
Pain (General disorders) | 3 | 11
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9 | 6
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 18 | 12
Peripheral sensory neuropathy (Nervous system disorders) | 7 | 3
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 | 0
Platelet count decreased (Investigations) | 22 | 12
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 8 | 7
Rectal hemorrhage (Gastrointestinal disorders) | 1 | 2
Renal and urinary disorders - Other (Renal and urinary disorders) | 2 | 0
Serum amylase increased (Investigations) | 0 | 3
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Sinusitis (Infections and infestations) | 4 | 0
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 1 | 4
Skin infection (Infections and infestations) | 2 | 1
Toothache (Gastrointestinal disorders) | 2 | 0
Upper respiratory infection (Infections and infestations) | 3 | 0
Urinary tract infection (Infections and infestations) | 2 | 0
Vascular disorders - Other (Vascular disorders) | 0 | 2
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Vomiting (Gastrointestinal disorders) | 14 | 3
Weight loss (Investigations) | 3 | 3
White blood cell decreased (Investigations) | 30 | 19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less